CLINICAL TRIAL: NCT04168463
Title: Exploring Use of Companion Robot Pets for Older Adults in Care Homes, an 8-month Stepped-wedge, Cluster Randomised Control Trial.
Brief Title: Exploring Use of Companion Robot Pets for Older Adults in Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Hannah Bradwell, Principal Investigator, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 268571
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Aging; Dementia; Neuropsychiatric Symptoms; Wellbeing
Keywords: Dementia; Social robots; Companion robots; Robot pets; Wellbeing; Older adults; Long-term care; Residential care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, cluster randomised control trial
Masking Description: N/A not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): This cluster of four homes will receive robot animals immediately at commencement of the eight month trial.
  Interventions: Device: Two Joy for All robots (one cat and one dog)
- Delayed Intervention (Other): This cluster of four homes will receive robot animals four months after commencement of the 8 month trial. The four months without robots will serve as a control period.
  Interventions: Device: Two Joy for All robots (one cat and one dog)

INTERVENTIONS:
Device: Two Joy for All robots (one cat and one dog) — Intervention will include the opportunity to interact with the Joy for All robot animals.
  Other Names: Robot pets; Companion robots

SUMMARY:
This study will assess the use and impact of the affordable 'Joy for All' robot pets for older people with and without dementia living in the care homes in South West England.

Robot pets such as Paro have shown potential in improving wellbeing (including reduced agitation, loneliness, medication use, anxiety and depression), however previous work conducted by the investigators suggests Paro is less acceptable to older adults than alternative devices; the Joy for All cat and dog. Paro is also much more expensive (£5000 compared to £100) limiting its use within the real world, and limiting the number of people able to benefit.

The investigators therefore wish to explore the potential of these more affordable robots in achieving wellbeing benefits.

DETAILED DESCRIPTION:
This study will be an eight month stepped-wedge, cluster randomised control trial exploring the use and impact of 'Joy for All' robot pets with older people living in care homes in South West England. Participants will include individuals with and without dementia.

The study aims to:

* See if affordable robot pets lead to improved wellbeing and are robust and engaging over 4-8 months in care homes and nursing homes.
* Identify under what circumstances, for which care home residents, and with what impact the robot pets are used.

The wellbeing outcomes to be explored include; neuropsychiatric symptoms, challenging behaviour, communication and loneliness.

Additional outcomes include monitoring of medication use, 1:1 care applications, and maintenance of a usage chart.

Qualitative data will also be collected through reflective diaries maintained by care staff, and interviews following completion of the study.

The study will include residents of eight care homes, which will be stratified into two clusters based on size and dementia service. The two clusters will then be randomised to immediate start (and receive robot animals immediately), or delayed start (and receive robot animals after four months). This provides a period of control. The sample size is primarily informed by feasibility, and the number of residents in each home likely to participate. In total there are approximately 190 residents of which the investigators estimate 100 across the 8 homes will give consent and interact with the robots. If 70% residents (across both arms and over the whole study) benefit from interacting with the robots the 95% confidence interval is 61-79%. This is of sufficient precision.

Measures will be completed at baseline, 4 months and 8 months. Interviews will be conducted at 8 months, and analysed alongside reflective diary entries.

This study should provide understanding of the potential for these more affordable robot pets in improving wellbeing for older people, and insight into their use and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Any resident at a collaborating care home or nursing home that has consent to participate.

Exclusion Criteria:

* Any resident at a collaborating home without consent to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (Nursing Home Version) (Cummings, 1994) | Measured at baseline, 4 months and 8 months
  Will be used to assess any changes in neuropsychiatric symptoms of care home residents. For each domain, there are four scores; frequency (0-4, with higher scores being most frequent), severity (0-3, with higher scores being most severe), total score (frequency x severity), and caregiver distress (0-5, higher scores signal more distress)

SECONDARY OUTCOMES:
Challenging Behaviour Scale (Moniz-Cook et al., 2001) | Measured at baseline, 4 months and 8 months
  Will be used to assess any changes in challenging behaviour exhibited by care home residents. Scores range from 0-400, with higher scores indicating more challenging behaviours.
Campaign to End Loneliness Measurement Tool (3-item) (Campaign to End Loneliness, n.d.) | Measured at baseline, 4 months and 8 months
  Will be used to assess any changes in feelings of loneliness among care home residents. This outcome is measures with 3-items, scores range from 0-12, with higher scores indicating most loneliness.
Holden Communication Scale (Strøm et al., 2016) | Measured at baseline, 4 months and 8 months
  Will be used to assess any changes in communication of care home residents. Scores range from 0-48, with higher scores indicating more communication difficulties.
Medication Use Review | Will be reviewed for the 4 weeks prior to study commencement, 4 weeks prior to 4 month post study commencement and the 4 weeks prior to study completion at 8 months
  Medication charts will be reviewed to assess any changes in medication use, particularly anti-depressant or anti-psychotic or 'pro re nata' or PRN medications to alleviate mood or distress.
1:1 Care Applications | Will be reviewed for the 4 weeks prior to study commencement, 4 weeks prior to 4 month post study commencement and the 4 weeks prior to study completion at 8 months
  Will assess any changes in number of 1:1 care applications for each care home resident
Qualitative Impact Review | Dairies will be maintained during intervention phases (8 months for cluster 1, 4 months for cluster 2), interviews and summative review will be conducted at 8 months
  Review of diaries, staff interviews and staff summative review will allow qualitative assessment of impact that may have been missed on selected quantitative scales

CONTACTS AND LOCATIONS:
Overall Officials: Hannah L Bradwell, MSc, Principal Investigator — PhD Student, School of Nursing and Midwifery, University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moniz-Cook E, Woods R, Gardiner E, Silver M, Agar S. The Challenging Behaviour Scale (CBS): development of a scale for staff caring for older people in residential and nursing homes. Br J Clin Psychol. 2001 Sep;40(3):309-22. doi: 10.1348/014466501163715. PMID 11593958
- [Background] Strom BS, Engedal K, Saltyte Benth J, Grov EK. Psychometric evaluation of the Holden Communication Scale (HCS) for persons with dementia. BMJ Open. 2016 Dec 13;6(12):e013447. doi: 10.1136/bmjopen-2016-013447. PMID 27965255
- [Derived] Bradwell H, Edwards KJ, Winnington R, Thill S, Allgar V, Jones RB. Implementing Affordable Socially Assistive Pet Robots in Care Homes Before and During the COVID-19 Pandemic: Stratified Cluster Randomized Controlled Trial and Mixed Methods Study. JMIR Aging. 2022 Aug 24;5(3):e38864. doi: 10.2196/38864. PMID 35830959
- See also: Campaign to End Loneliness (n.d.) — https://www.campaigntoendloneliness.org/wp-content/uploads/Loneliness-Measurement-Guidance1-1.pdf
- See also: Holden Communication Scale — https://mafiadoc.com/the-holden-communication-scale-hcs_5a0b796c1723dd1abb6a85cb.html